CLINICAL TRIAL: NCT06400134
Title: Investigation of the Relationship of Cognitive Functions With Physical Performance, Grip Strength, Walking Speed, Mobility, and Frailty in Geriatric Individuals
Brief Title: Coginitve and Physical Functions in Geriatric İndividuals
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-08
Record Dates: First submitted 2024-04-30; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Cognitive Change; Physical Performance; Frailty; Mobility
MeSH Terms: conditions — Frailty | interventions — Neuropsychological Tests; Physical Functional Performance; Hand Strength; Walking Speed; Range of Motion, Articular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Geriatric individuals: Volunteer healthy geriatric individuals aged 65 years and over
  Interventions: Other: Cognitive Function; Other: Physical Performance; Other: Grip Strength; Other: Walking speed; Other: Mobility; Other: Fraility

INTERVENTIONS:
Other: Cognitive Function — The Standardized Mini Mental Test (SMMT) was used to evaluate the cognitive status of the geriatric individuals'. In the test, which has a total score of 30, those with a score of 24 or less are recommended to be evaluated for dementia.
Other: Physical Performance — The Brief Physical Performance Battery (BPPB) was used to assess the physical performance of geriatric individuals. All three physical performance measures (balance, walking speed, getting up from the chair) were scored between 0-4 according to the duration of the activity, these scores were summed and the total score was determined between 0 (poor) and 12 (very good).
Other: Grip Strength — Muscle strength was assessed with a hand grip dynamometer. In the geriatric individuals, less than 30 kg for men and less than 20 kg for women was considered as low hand grip strength.
Other: Walking speed — Walking speed was assessed with the 6-metre walk test. Speed was calculated by dividing each known distance by the time it took for each individual, on each trial, to walk from the start to the end points marked on the floor and then converting to m/s.
Other: Mobility — The Time up Go test (TUG) was used for mobility. The risk of falling increases with increasing duration.
Other: Fraility — Frailty assessment was performed using the FRAIL scale.The scale was scored by giving 0 or 1 point according to the answer given. The higher the score, the greater the fraility.

SUMMARY:
The aim of this study is to investigate the relationship between cognitive functions with physical performance, grip strength, walking speed, mobility, and frailty in geriatric individuals.

Decline in cognitive function and decline in physical performance are generally associated with advanced age. Cognitive dysfunction is a natural consequence of ageing and is an important factor in maintaining quality of life and independence. Investigating the relationship between cognition, physical performance, mobility, and frailty has become a challenging issue in recent years. However, there is a need to further clarify the direction of this cognitive-motor link.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer healthy geriatric individuals aged 65 years and over
* Able to walk independently

Exclusion Criteria:

* Without neurological and rheumatological diseases,
* Without acute musculoskeletal problems in the lower extremities

Ages: 65 Years to 82 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Geriatric individuals
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Cognition function | 4 month
  The Standardised Mini Mental Test, which evaluates cognitive functions, consists of a total of 30 points. Those who score 24 and below are evaluated for dementia.

SECONDARY OUTCOMES:
Physical Performance | 4 month
  The Brief Physical Performance Battery (BPPB) was used to assess the physical performance.All three physical performance measures (balance, walking speed, getting up from the chair) were scored between 0-4 according to the duration of the activity, these scores were summed and the total score was determined between 0 (poor) and 12 (very good).
Grip Strength | 4 month
  Muscle strength was assessed with a hand grip dynamometer. In the geriatric individuals, less than 30 kg for men and less than 20 kg for women was considered as low hand grip strength
Walking speed | 1 month
  Walking speed was assessed with the 6-metre walk test. Speed was calculated by dividing each known distance by the time it took for each individual, on each trial, to walk from the start to the end points marked on the floor and then converting to m/s
Mobility | 4 month
  The Time up Go test (TUG) was used for mobility. Completion in more than 12 seconds indicates a high fall risk in geriatric individuals
Frailty | 4 month
  Frailty assessment was performed using the FRAIL scale. The scale was scored by giving 0 or 1 point according to the answer given. As a result, a total score of 0 was defined as normal, between 1-2 points as pre-frailty, and above 2 points as frail

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Ankara Yıldırım Beyazıt University, Faculty of Health Sciences,Department of Physiotherapy and Rehabilitation, Ankara, Esenboğa
  - Ankara Yıldırım Beyazıt University, Ankara